CLINICAL TRIAL: NCT01464814
Title: A Double Blind Placebo Controlled Crossover Clinical Trial Evaluating The Viability Of KE-99 With Fish Oil In Healthy Adults
Brief Title: Clinical Trial Evaluating the Viability of L. Casei + Fish Oil Capsules
Acronym: Probiomega
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nutrition 21, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: N21-2011
Record Dates: First submitted 2011-10-04; First posted 2011-11-04 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Signs and Symptoms, Digestive
Keywords: probiotic; fish oil; digestion; viability
MeSH Terms: conditions — Signs and Symptoms, Digestive | interventions — Probiotics; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Experimental): Lactobacillus casei in fish oil capsule
  Interventions: Dietary Supplement: probiotic plus fish oil capsule
- Placebo (Placebo Comparator): Fish oil capsule
  Interventions: Dietary Supplement: Fish oil capsule

INTERVENTIONS:
Dietary Supplement: probiotic plus fish oil capsule — Lactobacillus casei (4B CFU) plus fish oil capsule, T.I.D., for seven (7) days.
  Other Names: Probiomega
  Arms: Probiotic
Dietary Supplement: Fish oil capsule — Fish oil capsule, T.I.D., for seven (7) days
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effects of the probiotic KE-99 Lactobacillus casei when administered with omega-3 fish oil on probiotic viability, fecal make-up and gastrointestinal (GI) health in healthy adults.

DETAILED DESCRIPTION:
This is a randomized, placebo controlled, crossover clinical trial to determine the effects of KE-99 Lactobacillus casei with omega-3 fish oil, a probiotic purported to promote beneficial effects in gastrointestinal (GI) health. The study will last approximately three weeks with subjects attending a screening visit and four follow-up visits.

The study will involve subjects taking the probiotic product (KE-99 + fish oil)and placebo, each for seven days (as per sponsor guidance), in random order, with a seven day washout in between (as per sponsor guidance). Fecal analyses will be done at the beginning and end of each seven day supplementation period so that the number of live KE-99 in feces can be determined with higher numbers being positive (indicates more live KE-99 survived digestion).

Although the study population will be comprised of generally healthy adults that do not have GI disorders or symptoms, the sponsor hypothesizes that there may be beneficial effects in GI health with the KE-99 + fish oil supplementation. A six item questionnaire will be used to assess changes in GI health (e.g. abdominal pain, bloating and gas) with lower incidence indicating positive effects with regard to GI health.

ELIGIBILITY:
Inclusion Criteria:

* Female subject is surgically sterile, post-menopausal or agrees to use an acceptable method of birth control
* Subject is able to understand and sign the informed consent to participate in the study
* Subject is willing and able to comply with the protocol including:a. Attending five visits; b. Collecting four stool samples; c. Refraining from eating any yogurt or lacto-fermented beverages during the study; d. Refraining from using any dietary supplements including probiotics or prebiotics during the study;e. Not taking any new vitamin and/or mineral supplements until after study completion.

Exclusion Criteria:

* Subject has any of the following medical conditions: a. active heart disease, b. uncontrolled high blood pressure (≥ 140/90 mmHg), c. renal or hepatic impairment/disease, d. Type I or II diabetes, e. bipolar disorder f. Parkinson's disease, g. unstable thyroid disease, h. immune disorder (such as HIV/AIDS), i. psychiatric disorders (hospitalized within the past one year), j. any medical condition deemed exclusionary by the Principal Investigator (PI)
* Subject has a history of cancer (except localized skin cancer without metastases or in situ cervical cancer) within five years prior to screening.
* Subject has a history of or currently has any gastrointestinal disease or disorder or any inflammatory bowel condition such as Crohn's disease, short bowel,ulcerative colitis, or Irritable Bowel Syndrome (IBS).
* Subject has constipation defined as less than three spontaneous bowel movements per week.
* Subject is lactose intolerant (self-professed or diagnosed).
* Subject has had any stomach or intestinal surgery (i.e. gastric bypass).
* Subject takes on a regular basis (defined as two or more times per week) any prescription or over-the counter medications for diarrhea, constipation, heartburn or any other gastrointestinal problems.
* Subject is currently taking laxatives or has taken laxatives within the 30 days prior to screening/enrollment.
* Subject is currently taking antibiotics (or any drug that significantly interferes with bacterial flora) or has taken antibiotics within the 60 days prior to screening/enrollment.
* Subject is currently taking or has used in the past 30 days probiotics (including yogurt and lacto-fermented beverages), prebiotic supplements, or any digestive enzymes [prescription or over-the-counter (OTC)]. Thirty-day washout allowed.
* Subject is on an unstable dose of medication (defined as fewer than 90 days at the same dose).
* Anti-hypertensives and anti-hyperlipidemic medications ok if stable dose.
* Subject is currently taking any medication deemed exclusionary by PI.
* Subject exhibits evidence of hepatic or renal dysfunction as evidenced by ALT, AST, AP being ≥ two times the upper limit of normal or serum creatinine value ≥ 2.0 mg/dl or other clinically significant abnormal clinical laboratory value per PI discretion.
* Subject has an allergy to fish or any of the ingredients in the test product (see section 3.2.1).
* Subject has a history of drug or alcohol abuse in the past 12 months.
* Subject has any condition or abnormality that, in the opinion of the investigator, would compromise the safety of the subject or the quality of the study data.
* Subject is participating or has participated in another research study within 30 days prior to the screening visit.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2011-10; Primary Completion 2011-11 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Fecal probiotic (KE-99) level | Fecal samples collected at baseline and after 7 days of treatment, during each treatment arm.
  KE-99 probiotic levels will be measured from fecal samples at baseline and compared to levels measured after 7 days of treatment to determine if live KE-99 bacteria survive transit through the gastrointestinal tract.

SECONDARY OUTCOMES:
SF-36v2 | At baseline and after 7 days of each treatment arm.
  SF-36v2 - is a multi-purpose, short-form health survey with 36 questions. It yields an 8-scale profile of functional health and well-being scores as well as psychometrically-based physical and mental health summary measures and a preference-based health utility index. Results will be compared between and within groups.
GI questionnaire | At baseline and after 7 days of each treatment arm.
  GI Questionnaire - a six-part questionnaire regarding general well-being and gastrointestinal symptoms will be administered, with results being compared between and within groups.
Tolerability Questionnaire | After 7 days of each treatment arm.
  Tolerability of the study products will be assessed at the end of each seven-day supplementation period (at visits 3 and 5).
qPCR Fecal Microbiota Analyses | Measuerd at baseline (Day 0) and after 7 days, of each treatment arm.
  Reverse transcription-quantitative PCR (RT-qPCR) will be performed at baseline (Day 0) and after 7 days of treatment, to compare human intestinal microbiota after treatment to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: David Seiden, MD, Principal Investigator — Broward Research Group
Locations (1):
- Broward Research Group, Pembroke Pines, Florida, United States